CLINICAL TRIAL: NCT06620731
Title: Single-dose, Parallel, Open-label Pharmacokinetic Study of FCN-437c Capsule in Subjects With Impaired Liver Function
Brief Title: Clinical Trial of FCN-437c Capsule in Patients With Hepatic Insufficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ahon Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FCN-437c-CP-005
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Hepatic Insufficiency
Keywords: Clinical Pharmacology; Hepatic insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — FCN-437c

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mild hepatic impairment group (Experimental): participants with mild hepatic impairment(Child-Pugh A)
  Interventions: Drug: FCN-437c capsule
- moderate hepatic impairment group (Experimental): participants with moderate hepatic impairment (Child-Pugh B)
  Interventions: Drug: FCN-437c capsule
- health volunteer group (Experimental): Normal hepatic function
  Interventions: Drug: FCN-437c capsule

INTERVENTIONS:
Drug: FCN-437c capsule — Take 200 mg of FCN-437c capsules with approximately 240 mL of warm water in the morning on an empty stomach.

SUMMARY:
To evaluate and compare the safety and efficacy of FCN-437c in subjects with mild and moderate liver impairment and healthy subjects, and to provide a basis for clinical medication in patients with liver impairment.

ELIGIBILITY:
Inclusion Criteria:

Subjects with hepatic impairment must meet all of the following criteria to enter this study.

1. Sign the informed consent form before the trial, and fully understand the content, process and possible adverse effects of the trial, and be willing to strictly comply with the requirements of the trial program to complete the study.
2. 18 to 75 years of age (both sexes) on the date of signing the informed consent form.
3. Males weighing ≥ 50 kg, females weighing ≥ 45 kg, with a body mass index (BMI) in the range of 18 kg/m 2 ~32 kg/m 2 (including threshold values).
4. Chronic, stable (no clinically significant change in disease status prior to study drug administration, as determined by the investigator), hepatic impairment due to primary liver disease (e.g., hepatitis B, hepatitis C, autoimmune hepatitis, non-alcoholic fatty liver disease, alcoholic liver disease, etc.), assessed as Grade A/mild (Child-Pugh score: 5-6) or Grade B/moderate (Child-Pugh score: 7-9) prior to study drug administration; in which the investigator uses standardized diagnostic techniques, the investigator uses standard diagnostic techniques, and the investigator uses standardized treatment methods to determine whether the disease is clinically stable or clinically stable. Those who have Grade A/mild (Child-Pugh Score: 5-6) or Grade B/moderate (Child-Pugh Score: 7-9) liver dysfunction; among them, those who are diagnosed with chronic liver dysfunction by the investigator using standardized diagnostic methods, combined with the patient's past medical history, laboratory tests, liver biopsy, or imaging studies, etc. will be evaluated according to the Child-Pugh Score;
5. have had a stable regimen of medications for hepatic impairment, complications, and other concomitant conditions for at least 14 days prior to administration of study drug, which does not require adjustment of the medication (including type of medication, dosage, or frequency of medication) (except for subjects with moderate hepatic impairment who require the use of an oral diuretic at any time if ascites is present); or have not been on medication.
6. Vital organ function meets the following criteria.

   * Neutrophil count (ANC) ≥1.0 x 10 9 /L (1,000/mm 3 ).
   * Platelets ≥ 50.0 x 10 9 /L (50,000/mm 3 ).
   * Hemoglobin (Hgb) ≥7.0 g/dL (70 g/L).
   * Albuminous aminotransferase (ALT) and albuminous aminotransferase (AST) ≤ 5 times the upper limit of normal (ULN);
   * Creatinine clearance (CLcr, calculated using the Cockcroft-Gault formula for creatinine clearance, Annex II) > 60mL/min.
   * QTc interval (QTcF) corrected by Fridericia's criteria ≤470 msec in men and ≤480 msec in women.
7. The investigator determines the acceptable physical status based on the subject's medical history, physical examination, vital signs, laboratory tests (routine blood, blood biochemistry, urinalysis, coagulation, etc.), and 12-lead electrocardiogram;
8. Male and female subjects of childbearing potential are willing to use adequate and effective contraception after signing the informed consent form, during the study, and for 6 months after administration of study medication; women of childbearing potential must have a negative serum pregnancy test within 24 days prior to study drug administration.

Healthy subjects must meet all of the following criteria to enter this study.

1. Sign the informed consent form before the trial, and fully understand the content, process and possible adverse effects of the trial, and be willing to strictly comply with the requirements of the trial program to complete the study.
2. On the date of signing the informed consent form, the patients were 18 to 75 years old (including both ends)(required age matching with the liver function impairment group, the average age of the healthy subjects group was within the range of the average age of the mild and moderate liver function impairment group ±10 years), both men and women (required gender matching with the liver function impairment group, the average age of the liver function impairment group was within the range of the liver function impairment group ±10 years). The number of subjects per sex in the healthy group was required to be similar to that in the mild and moderate liver dysfunction groups (±1 subject/sex).
3. Male weight ≥ 50 kg, female weight ≥ 45 kg, body mass index (BMI) within the range of 18 kg/m 2 ~32 kg/m 2 (including the threshold value) (to be weight-matched with the hepatic impairment group, the average weight of the healthy subjects group is within the range of the average weight of the group with mild and moderate hepatic impairment ± 10 kg).
4. Normal or abnormal physical examination, vital signs, laboratory tests (blood, blood biochemistry, urine, prothrombin, etc.), 12-lead electrocardiogram, abdominal ultrasound, etc. that are not clinically significant in the judgment of the investigator.
5. Male and female subjects of childbearing potential are willing to use adequate and effective contraception after signing the informed consent form, during the study period, and for 6 months after taking the study drug; women of childbearing potential must have had a negative serum pregnancy test within 24 h prior to the administration of study drug.

Exclusion Criteria:

Subjects with hepatic impairment will be excluded from the study if they meet any of the following criteria.

1. Subjects with any of the following conditions: drug induced liver injury; history of liver transplantation; cirrhotic patients with liver failure or complications such as grade 3/4 hepatic encephalopathy, ruptured varices of the fundus esophagus, or hemorrhage, which in the opinion of the investigator are inappropriate; severe/advanced peritoneal or pleural effusions requiring puncture drainage and albumin supplementation.
2. Diseases affecting the excretion of bile, such as biliary cirrhosis.
3. those with severe portal hypertension or previous portosystemic shunts, including transjugular intrahepatic portosystemic shunts.
4. In addition to primary diseases of the liver, have previously suffered from serious primary diseases of other important organs, including but not limited to neuropsychiatric, gastrointestinal, respiratory, urinary, endocrine, hematological, immunological, etc., which, in the judgment of the investigator, make them unsuitable for participation in this trial.
5. Myocardial infarction, severe/unstable colic, symptomatic congestive heart failure (NYHA class II-IV), or clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention within 6 months prior to study entry.
6. any other malignancy diagnosed within 5 years prior to study participation, except for radically treated early stage malignancies (carcinoma in situ or stage I tumors), such as adequately treated basal cell or squamous cell skin cancers or carcinoma in situ of the cervix.
7. severe infection, trauma, gastrointestinal surgery or other major surgical procedure within 4 weeks prior to screening;
8. have lost or donated ≥400 mL of blood or received a red blood cell transfusion within 1 month prior to screening; or have taken any clinical trial medication within 1 month prior to screening.
9. allergy, including a history of severe drug allergy or drug metabolism; known hypersensitivity to FCN-437C capsule or its excipients.
10. Regular drinkers (≥14 units of alcohol per week: 1 unit = 360 mL of beer, or 45 mL of 40% alcohol by volume, or 150 mL of wine) in the 6 months prior to screening; smokers ≥5 cigarettes per day in the 3 months prior to screening; those with a positive alcohol screen; and those who are unable to abstain from smoking and alcohol for the duration of the trial.
11. a history of drug use, or a history of substance abuse within the past 5 years, or a positive drug screen (except for a positive drug screen due to concomitant medication use).
12. HIV antibody-positive and syphilis antibody-positive patients; syphilis antibody-positive patients can be enrolled if they are negative for RPR.
13. pregnant or breastfeeding women.
14. persons who have received a live (attenuated) vaccine (other than influenza vaccine) within 14 days prior to screening or who plan to receive it during the course of the trial.
15. who have taken a strong or moderate inducer or strong or moderate inhibitor of CYP3A (Annex III), or prescription, over-the-counter, herbal, or dietary supplements other than medications for the treatment of hepatic impairment and other concomitant diseases within 14 days prior to administration of study drug.
16. ingestion of grapefruit or grapefruit-containing products, fruit juices, foods or beverages containing methylxanthines (e.g., tea, coffee, cola, chocolate, functional beverages) or alcohol within 72 hours prior to the administration of the study drug; strenuous physical activity; or any other factor that affects the absorption, distribution, metabolism, excretion, etc. of the drug.
17. the presence of other serious physical or mental illnesses or abnormal laboratory tests, and other factors that may increase the risk of participation in the study or interfere with the results of the study; and any other condition that, in the opinion of the investigator, makes participation in this study inappropriate.

Healthy subjects were not eligible to participate in this study if they met any of the following criteria.

1. a previous history of liver impairment, or a physical examination and laboratory tests at the time of screening suggesting the presence or potential presence of liver impairment.
2. Previously suffered from primary diseases of important organs, including but not limited to neuropsychiatric, cardiovascular, gastrointestinal, respiratory, urinary, endocrine, hematological, immunological, etc., which, in the judgment of the investigator, are not suitable for participation in this trial;
3. severe infection, trauma, gastrointestinal surgery or other major surgical procedure within 4 weeks prior to screening;
4. have lost or donated ≥400 mL of blood or received a blood transfusion within 3 months prior to screening; or have taken any clinical trial medication.
5. allergy, including a history of severe drug allergy or drug metabolism; known hypersensitivity to FCN-437c capsule or its excipients.
6. Regular alcohol drinkers in the 6 months prior to screening (≥14 units of alcohol per week: 1 unit=beer 360 mL, or 45 mL of 40% alcohol by volume spirits, or 150 mL of wine); smoked ≥5 cigarettes per day in the 3 months prior to screening; screened positive for alcohol; and were unable to abstain from smoking and alcohol during the trial.
7. a history of drug abuse, or a history of substance abuse within the past five years, or a positive drug screen.
8. Hepatitis B surface antigen (HBsAg) positive, Hepatitis C (HCV) antibody positive, HIV antibody positive, Syphilis antibody positive.
9. QTc intervals (QTcF) corrected by Fridericia's criteria >470 msec in men and >480 msec in women.
10. pregnant or breastfeeding women.
11. persons who have received a live attenuated vaccine within 14 days prior to screening or who plan to receive a vaccine during the course of the trial (except for influenza vaccine).
12. have taken an inducer or inhibitor of CYP3A (Annex III), or any prescription, over-the-counter, herbal, or dietary supplement within 14 days prior to administration of study drug.
13. ingestion of grapefruit or grapefruit-containing products, fruit juices, foods or beverages containing methylxanthines (e.g., tea, coffee, cola, chocolate, functional beverages) or alcohol within 72 hours prior to the administration of the study drug; strenuous physical activity; or any other factor that affects the absorption, distribution, metabolism, excretion, etc. of the drug.
14. the presence of other serious physical or mental illnesses or abnormal laboratory tests, and other factors that may increase the risk of participation in the study or interfere with the results of the study; and any other condition that, in the opinion of the investigator, makes participation in the study unsuitable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Cmax | Within 0.5 hours before administration to 192 hours after administration
  According to different liver function group measurement
AUC0-t | Within 0.5 hours before administration to 192 hours after administration
  According to different liver function group measurement
AUC0-∞ | Within 0.5 hours before administration to 192 hours after administration
  According to different liver function group measurement

SECONDARY OUTCOMES:
Tmax | Within 0.5 hours before administration to 192 hours after administration
  According to different liver function group measurement
t1/2 | Within 0.5 hours before administration to 192 hours after administration
  According to different liver function group measurement
CL/F | Within 0.5 hours before administration to 192 hours after administration
  According to different liver function group measurement
Vz/F | Within 0.5 hours before administration to 192 hours after administration
  According to different liver function group measurement
Fu | Within 0.5 hours before administration to 192 hours after administration
  According to different liver function group measurement
AUC0-t,u | Within 0.5 hours before administration to 192 hours after administration
  According to different liver function group measurement

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, PI, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu J, Liu J, Ding Y, Yang X, Fu Y, Sun Y. Safety and pharmacokinetics of FCN-437c, a novel cyclin-dependent kinase 4/6 inhibitor, in Chinese patients with hepatic impairment. Invest New Drugs. 2025 Aug;43(4):792-799. doi: 10.1007/s10637-025-01552-5. Epub 2025 Jul 15. PMID 40663244